CLINICAL TRIAL: NCT04306341
Title: Measuring the Impact of Real Time fMRI Neurofeedback in Borderline Personality Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: AE Foundation (Other); Central Institute of Mental Health, Mannheim (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000026750
Record Dates: First submitted 2020-03-10; First posted 2020-03-12 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Borderline Personality Disorder
MeSH Terms: conditions — Borderline Personality Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Neurofeedback in conjunction with Dialectical Behavior Therapy
  Interventions: Behavioral: real time fMRI neurofeedback
- Control (No Intervention): Dialectical Behavior Therapy (treatment as usual)

INTERVENTIONS:
Behavioral: real time fMRI neurofeedback — Participants will use real time feedback about their amygdala activity to learn to decrease amygdala activity.
  Arms: Experimental

SUMMARY:
This study will test the impacts of real time fMRI neurofeedback in patients with Borderline Personality Disorder. This is a pilot study in a small number of people enrolled in clinical programs at Yale New Haven Hospital.

ELIGIBILITY:
Inclusion Criteria:

1. enrolled in YNHH DBT-IOP
2. must meet specific clinical criteria
3. Inclusion in Experimental group requires participants meet standard safety and quality control requirements for MR scanning
4. For female participants, not pregnant and willing to use a reliable method of contraception during the study

Exclusion Criteria:

1. IQ<70
2. vision problem not able to be corrected to normal range
3. medication changes w/in one month
4. Lifetime hx of schizophrenia, schizoaffective d/o, bipolar I disorder.
5. illicit substance use within 7 days of MRI scans
6. taking scheduled opiates
7. taking scheduled benzodiazepines
8. taking scheduled anti-histamines
9. history of seizures
10. significant current or past neurologic illness
11. BMI < 16.5

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2020-11-15 (Actual); Primary Completion 2022-10-07 (Actual); Study Completion 2022-10-07 (Actual)

PRIMARY OUTCOMES:
Change in Affective Lability | Baseline compared to the week after intervention
  This outcome will be measured by the change in variance of negative emotions measured using ecologic momentary assessment (EMA: surveys sent to participants by smartphone app) repeatedly over a four-day period at each timepoint. The variance between measurements at each timepoint will be calculated, and compared to the other timepoints. There will be 5 negative emotion items at each timepoint, and a higher score indicates more negative emotion.

SECONDARY OUTCOMES:
Change in Mean Negative Affect | Baseline compared to the week after intervention
  This outcome will be measured by change in mean negative emotion score measured using ecologic momentary assessment (EMA: surveys sent to participants by smartphone app) repeatedly over a four-day period at each timepoint. The mean score at each timepoint will be calculated, and compared to the other timepoints. There will be 5 negative emotion items at each timepoint, and a higher score indicates more negative emotion.
Change in Borderline Personality Disorder Symptoms | Baseline compared to the week after intervention
  This outcome will be measured by change in Borderline Symptom List (BSL-23) score after neurofeedback. This scale has 23 items, each scored 0-4, and total score is mean item endorsement (sum of all items divided by 23). Higher scores indicate more symptom endorsement.
Change in Amygdala Regulation | Baseline compared to the week after intervention
  Change in ability to regulate amygdala activity when exposed to provocative images. Amygdala activity is measured as functional magnetic resonance imaging (fMRI) blood oxygen dependant (BOLD) signal

CONTACTS AND LOCATIONS:
Overall Officials: Sarah K Fineberg, MD PhD, Principal Investigator — Yale University; Michelle Hampson, PhD, Principal Investigator — Yale University
Locations (1):
- Connecticut Mental Health Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No